CLINICAL TRIAL: NCT02391558
Title: Clinical Evaluation of Noninvasive OCT Angiography Using a Zeiss OCT Prototype to Compare to Fluorescein Angiography
Acronym: OCTA
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: 4C-2015-07
Record Dates: First submitted 2015-03-12; First posted 2015-03-18 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Clinical evaluation of noninvasive OCT Angiography using a Zeiss OCT Prototype to replace fluorescein angiography.

DETAILED DESCRIPTION:
Fluorescein angiography (FA) is the standard and generally accepted method to identify vascular features in the retina, detecting capillary dropout and neovessel growth. Its value is undeniable and is a routine ophthalmological examination. However, it requires intravenous injection of fluorescein, which can cause nausea, vomiting and, rarely, anaphylaxis and death. New OCT angiography methods can detect, noninvasively red blood cells flow and, therefore, identify well the retinal vasculature. It is crucial and of major interest to evaluate the clinical utility of this new methodology comparing this information with the one obtained from fluorescein angiography.

ELIGIBILITY:
Inclusion Criteria:

* All patients with clinical indication for fluorescein angiography in their clinical practice

Exclusion Criteria:

* Subjects with a pacemaker of similarly critical electronic device
* Subjects with severe ocular media opacities
* Subjects with corneal abnormalities

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with clinical indication for fluorescein angiography will be invited to perform OCT angiography in the same day during a period of 6-8 months.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2015-09; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Comparison between examination techniques on the detection of morphological changes in the retina (such as vessels morphology, vascular ischemia, retinal neovascularization, choroidal neovascularization, and other vascular abnormalities). | Single Visit

CONTACTS AND LOCATIONS:
Locations (1):
- Aibili - Cec, Coimbra, Portugal

REFERENCES:
- [Derived] Soares M, Neves C, Marques IP, Pires I, Schwartz C, Costa MA, Santos T, Durbin M, Cunha-Vaz J. Comparison of diabetic retinopathy classification using fluorescein angiography and optical coherence tomography angiography. Br J Ophthalmol. 2017 Jan;101(1):62-68. doi: 10.1136/bjophthalmol-2016-309424. Epub 2016 Dec 7. PMID 27927677